CLINICAL TRIAL: NCT07328386
Title: Effect of Cervical Lymphaticovenous Anastomosis and Cervical Lymph Node to Vein Anastomosis for the Patient With Intracranial Lymphatic Circulation Disorder
Brief Title: Effect of Cervical Lymphaticovenous and Lymph Node-to-Vein Anastomosis in Patients With Intracranial Lymphatic Circulation Disorder
Acronym: CLVA-CLNA-ICLC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Joonpio (Other)
Responsible Party: Sponsor-Investigator, Hong Joonpio, Principal Investigator, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0033
Record Dates: First submitted 2025-11-25; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Intracranial Lymphatic Circulation Disorder; Alzheimer's Disease
Keywords: Lymphaticovenous Anastomosis (LVA); Lymph Node-to-Vein Anastomosis (LNVA); Amyloid Clearance; Cognitive Function; Dementia
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to one of two parallel groups:
  1. a surgical intervention group receiving cervical lymphaticovenous and lymph node-to-vein anastomosis plus standard medical therapy, and
  2. a control group receiving standard medical therapy alone. The two groups will be followed over the same time points to compare changes in cognitive and clinical outcomes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgical Intervention Group (Experimental): Participants in this group will undergo cervical lymphaticovenous anastomosis (LVA) and cervical lymph node-to-vein anastomosis (LNVA).
  The procedure connects cervical lymphatic vessels and lymph nodes to adjacent veins to facilitate lymphatic drainage from the brain and reduce amyloid accumulation associated with intracranial lymphatic circulation disorder in patients with Alzheimer's disease.
  Interventions: Procedure: Cervical Lymphaticovenous and Lymph Node-to-Vein Anastomosis
- Control Group (No Intervention): Participants in this group will receive standard medication therapy only, following the hospital's routine treatment guidelines for Alzheimer's disease.

INTERVENTIONS:
Procedure: Cervical Lymphaticovenous and Lymph Node-to-Vein Anastomosis — This microsurgical procedure involves connecting the cervical lymphatic vessels and lymph nodes to adjacent veins to enhance lymphatic drainage from the brain. The purpose of the surgery is to reduce amyloid accumulation and improve cognitive function in patients with intracranial lymphatic circulation disorders.
  Before the operation, ultrasound imaging is used to identify the lymphatic vessels, lymph nodes, and nearby veins. A small incision of approximately 2-3 cm is made along the sternocleidomastoid muscle. Indocyanine green (ICG) dye is injected to visualize lymphatic flow, and under microscopic guidance, the lymphatic structures are anastomosed to the adjacent veins. Finally, the incision is closed with adhesive, and no postoperative drainage is required.
  Arms: Surgical Intervention Group

SUMMARY:
This study is a single-center, prospective clinical trial designed to evaluate the therapeutic effects of lymphaticovenular anastomosis (LVA) and lymph node-venous anastomosis (LNVA) in patients with intracranial lymphatic circulation disorders. Following voluntary written informed consent, screening assessments will be performed in accordance with the clinical trial protocol. Eligibility will be determined based on the predefined inclusion and exclusion criteria, and eligible subjects will be enrolled in the study. Enrolled participants will undergo cognitive function assessments at baseline (pre-surgery) and at 1, 3, 6, 9, 12, 18, and 24 months postoperatively for follow-up. Cognitive evaluations will not be additionally performed for research purposes but will be conducted in accordance with the existing clinical care schedule and standard treatment guidelines.

DETAILED DESCRIPTION:
There are several theories regarding the causes of mild cognitive impairment (MCI) and dementia, and one of the commonly proposed mechanisms involves the accumulation of amyloid, a metabolic waste product, within the brain parenchyma. This accumulation is thought to result from impaired clearance of waste from the brain. Accordingly, impaired function of the brain's waste drainage system may contribute to the development of cognitive symptoms.

Because waste clearance from the brain occurs through lymphatic pathways, dysfunction of lymphatic circulation has been identified as an important contributing factor to MCI and dementia. However, due to the minute diameter of lymphatic vessels-typically less than 1 mm-direct therapeutic interventions targeting lymphatic function have long remained unexplored.

Recent advances in supermicrosurgical techniques have enabled procedures on lymphatic vessels as small as 0.2-0.3 mm, leading to the development of novel treatments for lymphatic circulation disorders. For example, patients with upper or lower extremity lymphedema, a representative condition of lymphatic dysfunction, have shown significant improvement following lymphaticovenular anastomosis (LVA) or lymph node-venous anastomosis (LNVA).

Lymphedema results from obstruction or damage to lymphatic pathways, causing the accumulation of lymphatic fluid in tissues. LVA and LNVA are microsurgical procedures that create new bypass routes by connecting lymphatic vessels or lymph nodes directly to adjacent veins, thereby allowing lymphatic fluid to drain into the venous system and re-enter systemic circulation. These procedures have been performed for more than two decades, with excellent therapeutic outcomes reported over the past five years. At Asan Medical Center, more than 100 such procedures are successfully performed annually.

Furthermore, based on the same principle applied in limb lymphedema, recent case-level studies have suggested that performing LVA or LNVA in lymphatic pathways or lymph nodes responsible for cerebral waste clearance may improve degenerative neurological conditions, including Alzheimer's disease. Based on this accumulated knowledge and surgical expertise, cervical lymphaticovenular anastomosis and cervical lymph node-venous anastomosis will be performed to connect lymphatic vessels and lymph nodes involved in cerebral lymphatic drainage to adjacent veins.

It is hypothesized that this procedure may help slow disease progression, preserve quality of life, and potentially improve cognitive function in patients with mild cognitive impairment or dementia.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 19 years or older who are diagnosed with intracranial lymphatic circulation disorder based on neurological evaluation.
* Global Deterioration Scale (GDS) score between 3 and 5 at screening.
* Diagnosis of Alzheimer's disease confirmed by amyloid PET-CT or CSF amyloid testing, showing amyloid accumulation associated with lymphatic circulation disorder.
* Able to provide written informed consent to participate in the study voluntarily.

Exclusion Criteria:

* Unable to undergo follow-up evaluation for at least 12 months after surgery.
* Diagnosed with vascular dementia.
* Presence of structural brain disease other than intracranial lymphatic circulation disorder.
* Known hypersensitivity to indocyanine green (ICG).
* Uncontrolled systemic medical conditions such as severe cardiopulmonary, renal, hepatic, or endocrine disorders.
* History of previous neck surgery.
* Refusal to participate or failure to provide informed consent.
* Determined by the principal investigator to be unsuitable for participation due to any other clinical reason.

Ages: 19 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Global Deterioration Scale (GDS) Score | From preoperative baseline to postoperative Months 1, 3, 6, 9, 12, 18, and 24
  Cognitive decline will be assessed using the Global Deterioration Scale (GDS). The GDS score ranges from 1 to 7, with higher scores indicating more severe cognitive impairment. The outcome measure is the change in GDS score from baseline to postoperative follow-up visits. Scores will be compared between the surgical (LVA + LNVA) group and the medication-only control group.
Change in Clinical Dementia Rating - Sum of Boxes (CDR-SB) Score | Preoperative baseline and postoperative Month 12
  Dementia severity will be evaluated using the Clinical Dementia Rating - Sum of Boxes (CDR-SB).
  CDR-SB scores range from 0 to 18, with higher scores indicating more severe cognitive impairment The outcome measure is the change in CDR-SB score from baseline to postoperative follow-up visits.
  Scores will be compared between the surgical (LVA + LNVA) group and the medication-only control group.
Change in Korean Mini-Mental State Examination (K-MMSE) Score | From preoperative baseline to postoperative Months 1, 3, 6, 9, 12, 18, and 24
  Cognitive function will be assessed using the Korean Mini-Mental State Examination (K-MMSE).
  K-MMSE scores range from 0 to 30, with higher scores indicating better cognitive function.
  The outcome measure is the change in K-MMSE scores from the preoperative baseline to 12 months after surgery.
  Scores will be compared between the surgical (LVA + LNVA) group and the medication-only control group.
Change in Montreal Cognitive Assessment (MoCA) Score | Preoperative baseline; postoperative Day 4; Months 1, 3, 6, 9, 12, 18, and 24
  Cognitive performance will be assessed using the Montreal Cognitive Assessment (MoCA).
  MoCA scores range from 0 to 30, with higher scores indicating better cognitive performance.
  The outcome measure is the change in MoCA scores from the preoperative baseline to 12 months after surgery.
  Scores will be compared between the surgical (LVA + LNVA) group and the medication-only control group.
Change in Seoul Neuropsychological Screening Battery (SNSB) Score | Preoperative baseline; postoperative Months 6, 12, and 24
  Cognitive function will be assessed using the Seoul Neuropsychological Screening Battery (SNSB), a comprehensive neuropsychological test battery evaluating multiple cognitive domains including attention, language, visuospatial function, memory, and executive function.
  SNSB provides domain-specific and composite scores, with higher scores generally indicating better cognitive performance, depending on the specific subtest.
  Score ranges differ across subtests within the SNSB. The outcome measure is the change in SNSB scores from the preoperative baseline to postoperative follow-up assessments.
  Scores will be compared between the surgical (LVA + LNVA) group and the medication-only control group.

SECONDARY OUTCOMES:
Incidence of Surgical Complications and Adverse Events | From the day of surgery through postoperative Month 24
  Surgical complications and adverse events will be monitored throughout the study period to evaluate the safety of cervical lymphaticovenous and lymph node-to-vein anastomosis.
  Complications may include postoperative infection, wound issues, bleeding, lymphatic leakage, anesthetic complications, or other procedure-related adverse events.
  Adverse events will be recorded according to clinical severity and temporal relationship to the intervention.
  The outcome measure is the incidence and type of complications occurring during the follow-up period.
Change in Amyloid-Related Blood Biomarkers | Preoperative baseline; postoperative Months 1, 3, 6, 12, and 24
  The outcome measure is the change from the preoperative baseline to postoperative follow-up assessments in pre-specified amyloid-related blood biomarkers (e.g., amyloid-beta-related markers). Changes in amyloid-related blood biomarkers will be compared between the surgical (LVA + LNVA) group and the medication-only control group.
Change in Blood Biomarkers of Neurodegeneration | Preoperative baseline; postoperative Months 1, 3, 6, 12, and 24
  The outcome measure is the change from the preoperative baseline to postoperative follow-up assessments in pre-specified blood biomarkers of neurodegeneration (e.g., phosphorylated tau). Changes in neurodegeneration-related blood biomarkers will be compared between the surgical (LVA + LNVA) group and the medication-only control group.

OTHER OUTCOMES:
Change in Gait Function Test Performance | Screening; postoperative Months 1, 3, 6, 9, 12, 18, and 24
  The outcome measure is the change in gait function from the screening assessment to postoperative follow-up assessments, as measured by a standardized gait function test yielding a single composite score according to the study protocol.
Change in Amyloid PET Imaging Findings | Screening; postoperative Month 6
  Amyloid positron emission tomography (PET) imaging will be performed to observe any changes in amyloid-related findings before and after the surgical intervention.
  PET imaging is conducted at screening to confirm eligibility and again at postoperative Month 6 to evaluate interval changes.
  Any differences in overall PET imaging appearance between the two time points will be examined and compared between the surgical (LVA + LNVA) group and the medication-only control group.

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No